CLINICAL TRIAL: NCT00155545
Title: Influence of Leg Length Discrepancy on the Spinal Shape and Biomechanics During Static and Dynamic Activities in Functional and Idiopathic Scoliosis Patients
Brief Title: Influence of Leg Length Discrepancy on the Spinal Shape and Biomechanics in Functional and Idiopathic Scoliosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 9361701286
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-11

CONDITIONS: Leg Length Discrepancy; Scoliosis
Keywords: functional scoliosis; idiopathic scoliosis; leg length discrepancy; motion analysis; biomechanics
MeSH Terms: conditions — Leg Length Inequality; Scoliosis

ARMS (1):
- Metformin (No Intervention)
  Interventions: Behavioral: Motion analysis of patients

INTERVENTIONS:
Behavioral: Motion analysis of patients

SUMMARY:
The purposes of this study are to use motion analysis techniques to study the biomechanical interactions between the spine and the lower limbs in scoliosis patients with or without leg length discrepancy (LLD) during activity; to investigate the effects of correction of LLD: using foot orthosis on the functional scoliotic spinal curve and motion during functional activity; and to test whether idiopathic scoliosis without LLD can be improved by artificially creating a leg length discrepancy with a foot orthosis.

DETAILED DESCRIPTION:
Scoliosis is one of the most common back deformities in children. Idiopathic and functional (secondary) scoliosis are arguably the two most common types. The etiology of idiopathic scoliosis has been studied in many aspects such as genetic factors, skeletal muscle abnormalities, neurological mechanisms, and biomechanical factors, while the common causes of secondary or functional scoliosis are leg length inequality and muscle spasm. It is evident that biomechanical factors that involve the interactions of the musculoskeletal alignment and loading are closely associated with the development of both types of scoliosis.

Leg length discrepancy (LLD) is defined as a condition in which paired limbs are unequal in length. It is now generally accepted that LLD can lead to lumbar scoliosis and it is assumed that scoliosis caused by LLD can be removed if LLD is eliminated. However, no study has documented the effects of the correction of LLD on the functional scoliotic spinal curve and motion during functional activity. Since spinal curve and motion have clear associations with leg length inequality, one would wonder whether idiopathic scoliosis without LLD can be improved by artificially creating a leg length difference with an orthosis when spine surgery is not considered or in a less severe condition. It has been shown that LLD and scoliosis have effects on pain, force transmission and performance of motion. Therefore, the artificially created leg length difference may have negative effects even though the scoliosis is improved. The benefits and disadvantages of using a foot orthosis to create artificial LLD in order to relieve idiopathic scoliosis require careful investigation. Although the biomechanics of the spine or the lower extremities have been studied separately in the literature, the biomechanical interactions between the spine and the lower limbs in scoliosis patients with or without LLD and the biomechanical effects of treatments using foot orthosis on these patients remain to be studied.

Using motion analysis techniques, the present study aims:

1. to study the biomechanical interactions between the spine and the lower limbs in scoliosis patients with or without LLD during activity;
2. to investigate effects of correction of LLD using a foot orthosis on the functional scoliotic spinal curve and motion during functional activity; and
3. to test whether idiopathic scoliosis without LLD can be improved by artificially creating a leg length discrepancy with a foot orthosis. The optimal heights of the foot orthosis for the later two objectives will also be determined. It is hoped that the present study will lead to a better understanding of the mechanical interactions between the spine and the lower extremities in functional and idiopathic scoliosis patients, and a better treatment for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Functional scoliosis patients who have lumbar scoliosis combined with significant structural LLD
* Adolescent idiopathic lumbar scoliosis patients without LLD

Exclusion Criteria:

* Do not suit the inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Variation of spine angle | 30
Variation of spine shape | 30

CONTACTS AND LOCATIONS:
Overall Officials: Shier-Chieg Huang, MD, Study Chair — Department of Orthopaedics, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan